CLINICAL TRIAL: NCT04905316
Title: Phase I/II Study of Canakinumab With Chemoradiation and Durvalumab for Unresected Locally-Advanced Non-Small Cell Lung Cancer (CHORUS)
Brief Title: A Study of Canakinumab With Chemotherapy, Radiation Therapy, and Durvalumab in People With Lung Cancer
Acronym: CHORUS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-004
Record Dates: First submitted 2021-05-24; First posted 2021-05-27 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Locally-advanced NSCLC (stage IIIA-C); Canakinumab; Durvalumab; Chemoradiation; 21-004
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — canakinumab; durvalumab; Radiotherapy; Drug Therapy

STUDY DESIGN:
Intervention Model Description: This is a single-arm, prospective, phase I/II study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Canakinumab with Chemoradiation and Durvalumab (Experimental): Treatment will consist of canakinumab (ACZ885) administered as a subcutaneous injection every 3 weeks for 3 cycles concurrent with standard of care concurrent chemoradiation, followed by canakinumab administered intravenously every 4 weeks for up to 12 total infusions concurrent with standard of care durvalumab. Canakinumab (ACZ885) will be dosed at 200mg via subcutaneous injection every 3 weeks x 3 injections that will start with concurrent chemoradiation, followed by 200mg via intravenous infusion every 4 weeks x 12 infusions that will start with the initiation of durvalumab. Canakinumab (ACZ885) will be concurrent with thoracic chemoradiation and durvalumab therapy for up to 15 cycles, or until disease progression or unacceptable toxicity, whichever occurs first. Patients that come off treatment for progression, or have progression after completion of all protocol-related therapy, can be followed for survival outcomes by chart review based on standard of care evaluations.
  Interventions: Drug: Canakinumab; Drug: Durvalumab; Radiation: Radiation therapy; Drug: Chemotherapy

INTERVENTIONS:
Drug: Canakinumab — Canakinumab (ACZ885) will be dosed at 200mg via subcutaneous injection every 3 weeks x 3 injections that will start with concurrent chemoradiation, followed by 200mg via intravenous infusion every 4 weeks x 12 infusions that will start with the initiation of durvalumab. Intravenous Canakinumab (ACZ885) should start no sooner than 3 weeks after the last subcutaneous Canakinumab (ACZ885) injection. Canakinumab (ACZ885) will be concurrent with thoracic chemoradiation and durvalumab therapy for up to 15 cycles, or until disease progression or unacceptable toxicity, whichever occurs first.
  Other Names: ACZ885
Drug: Durvalumab — Patients will be treated with durvalumab either at a dose of 10mg per kilogram of body weight intravenously every 2 weeks or at a 1500 mg fixed dose administered every 4 weeks as consolidation therapy after completion of concurrent chemoradiation therapy, as per standard of care.
Radiation: Radiation therapy — Radiation therapy will be performed with external beam ionizing radiation as per standard of care in accordance with institutional practice. Intensity-modulated radiation therapy (IMRT) or volumetric arc therapy (VMAT) will be used at the discretion of the treating radiation oncologist. Patients will be simulated in the treatment position with standard immobilization techniques for thoracic radiotherapy. The prescription dose will be 60 Gy (±10%) in 2Gy fractions to fields encompassing gross tumor and lymph nodes, as per institutional guidelines. The dose must satisfy institutional guidelines and minimize risk to adjacent organs at risk.
Drug: Chemotherapy — Chemotherapy will be as per standard of care in accordance with institutional practice. Patients will be treated with carboplatin or cisplatin with etoposide, paclitaxel, albumin-bound paclitaxel or pemetrexed at the discretion of the treating thoracic medical oncologist. Chemotherapy will be concurrent with radiation therapy as per standard practice, with cycle 1 day 1 of chemotherapy starting on fraction 1 of radiation ± 5 days.

SUMMARY:
The researchers are doing this study to find out whether canakinumab in combination with chemoradiation and durvalumab is an effective and safe treatment for people with locally advanced non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization obtained from the patient/legal representative prior to performing any protocol- related procedures, including screening evaluations.
* Patient age ≥ 18 at time of consent
* Stage IIIA-C NSCLC (as per the American Joint Commission on Cancer (AJCC) 8th edition)
* Not a candidate for surgical resection as determined by one or more of the following criteria in multidisciplinary evaluations: technically unresectable, medically inoperable, patient declines operative approach
* Candidate for concurrent chemoradiation therapy as determined by the treating radiation and thoracic oncologist
* Histologic confirmation of NSCLC with pathological review done at MSK
* ECOG Performance Status 0-1
* Candidate for definitive thoracic radiation (defined 60Gy ± 10% in 2 Gy fractions)
* Body weight > 30 kg
* Adequate normal organ and marrow function as defined below:

  * Hemoglobin ≥9.0 g/dL
  * Absolute neutrophil count (ANC) 1.5 x (> 1500 per mm3)
  * Platelet count ≥100 x 10^9/L (>100,000 per mm3)
  * Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
  * AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal
  * Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrhoeic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women <50 years of age would be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women ≥50 years of age would be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Must have a life expectancy of at least 6 months

Exclusion Criteria:

* Participation in another clinical study with an investigational (non-FDA approved) product during the last 4 weeks
* Concurrent enrollment in another clinical study for lung cancer, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
* Previous thoracic radiation precluding definitive RT
* Contraindication to Durvalumab
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients not on biologic therapy without active disease in the last 3 years may be included but only after consultation with the study physician
  * Patients with celiac disease controlled by diet alone
* Prior/Current Therapies:

  * Treatment with a administered > 4 weeks earlier (intraocular bevacizumab is acceptable).monoclonal antibody within 4 weeks prior to study Day 1 or has not recovered (i.e., ≥ Grade 1 at baseline) from adverse events due to agents
  * Patients receiving biologic drugs targeting the immune system (e.g. TNF blockers, anakinra, abatacept, tocilizumab) within 4 weeks prior to study Day 1
  * Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, anti-Cytotoxic Tlymphocyte-associated antigen-4 (CTLA-4) antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
  * Prior treatment with canakinumab
  * Current or prior use of a systemic immunosuppressive medication within 14 days before the first dose of canakinumab. The following are exceptions to this criterion:

    i. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection) ii. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent for less than 30 days. iii. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication) iv. Systemic glucocorticoid replacement for conditions such as adrenal or pituitary insufficiency.
* Major surgical procedure (e.g. intra-cranial, intra-thoracic, intra-abdominal, or intra-pelvic) within 28 days prior to the first dose of canakinumab
* Prior history of malignant disease, other than this NSCLC, that has been diagnosed and/or required therapy within the past 3 years. Exceptions to this exclusion include: completely resected basal cell and squamous cell skin cancers, completely resected carcinoma in situ of any type, and definitely treated Stage 0-I breast cancers on hormonal maintenance therapy or definitely treated Stage I-IIA prostate cancer.
* History of allogenic organ transplantation.
* Known severe concurrent illness:

  * Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
  * Active or recurrent hepatic disorders including cirrhosis, hepatitis B and C. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
  * Active tuberculosis infection (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice)
  * Human Immunodeficiency Virus (positive HIV 1/2 antibodies).
  * Active infection requiring systemic therapy.
  * Evidence of interstitial lung disease or active, non-infectious pneumonitis.
  * Clinically significant (i.e., active) cardiovascular disease: symptomatic cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential unless they are willing to employ a highly effective birth control from screening to 130 days after the last dose of canakinumab.

  °Highly effective methods of contraception, defined as one that results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly Note that condom use during intercourse among sexually actives males will be required. Note that some contraception methods are not considered highly effective (e.g. female cap, diaphragm, or sponge with or without spermicide; non-copper containing intrauterine device; progestogen-only oral hormonal contraceptive pills where inhibition of ovulation is not the primary mode of action [excluding Cerazette/desogestrel which is considered highly effective]; and triphasic combined oral contraceptive pills).
* Connective tissue disorders involving the lung(s) and/or esophagus requiring active treatment or idiopathic pulmonary fibrosis
* Known history of active primary immunodeficiency
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
* Receipt of live vaccination within 3 months prior to the first dose of study durg. Note that this only applies to live vaccines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 2 years

SECONDARY OUTCOMES:
Rate of grade ≥ 2 pneumonitis | 2 years
  by CTCAE v. 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Narek Shaverdian, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm